CLINICAL TRIAL: NCT06325917
Title: Effect of Self-management Education With Ongoing Support Using Social Media on Glycemic Control Among Patients With Diabetes Type 2.
Brief Title: Effect of Diabetes Self-management Education and Support on Glycemic Control Among Patients With Type 2 Diabetic
Acronym: DSMES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Jafar Alshraideh, Principal Investigator, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 101271-5
Record Dates: First submitted 2023-06-06; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Glycemic control; self-management education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: two arms parallel randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whatsApp ongoing support (Experimental): 70 patients will receive the usual care by DSN in the diabetes clinic through monthly visits supported by ongoing follow-up via what's App for a 3month.
  Interventions: Behavioral: what's app ongoing support
- usual care (Placebo Comparator): monthly follow-up at the diabetes education clinic patients receiving individual care and education by diabetes nurse specialist
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: what's app ongoing support — daily educational messages and reminders sent through WhatsApp. The educational material related to diabetes self-management behaviors (AADE7 Self-Care Behaviors, diabetes and genetics, and endocrinology center, also the Ministry of Health in Jordan diabetes.
  individual bidirectional communication between the participants and the investigator, which will allow participants to seek advice and get free-of-charge feedback and consultation.
  Arms: whatsApp ongoing support
Behavioral: usual care — monthly visit and follow-up at the diabetes education clinic by a diabetes nurse specialist providing DSMES
  Arms: usual care

SUMMARY:
Introduction: Diabetes mellitus (DM) is one of the chronic diseases that can have an impact on increasing morbidity, disability, and death. Social media has become a valuable resource for people with diabetes in improving self-management skills Applying diabetes self-management education with ongoing support using social media produces behavioral changes, empowerment, and cost-effectiveness.

purpose: the purpose of this study is to examine the effect of self-management education with ongoing support using social media (WhatsApp) on glycemic control among patients with uncontrolled diabetes.

Method: 140 patients with diabetes type 2 attending outpatients' diabetes clinic setting in Aqaba will participate in a two-arm randomized controlled trial study. Self-management education will be applied for all participants, ongoing support using social media (what's app) will be applied to the intervention group, and only usual diabetes care by a diabetes specialist nurse will be applied to the control group.

DETAILED DESCRIPTION:
Type 2 diabetes(DM2) consider a significant cause of morbidity and mortality worldwide. Around 1.5 million deaths globally, are directly attributed to diabetes each year. Adults with diabetes have a two- to three-fold increased risk of heart attacks and strokes, approximately, one million people were blinded due to diabetes. Also, Diabetes is the leading cause of kidney failure.

Uncontrolled DM2 has a negative impact on the healthcare system, patients, and community. Similarly, it has an adverse impact on the quality of life by its harmful complications that increase patients' disabilities, high hospitalization rates, and 30-day readmissions rate. Patients with DM2 have a high prevalence of DM-related stress. Additionally, a lack of diabetes awareness threatened patients' self-esteem stability, autonomy, and patient's ability to self-care and manage .

in Jordan, about 74.5 % of patients with DM had uncontrolled diabetes, despite their good knowledge level about diabetes and its complications. however, this knowledge did not translate into the ability to change patients 'behaviors regard to self-care activities this means that we need more innovative programs that encourage patients to utilize the knowledge they have .

Several unstructured diabetes self-management education (DSME) aimed to increase patients' awareness of the disease and its management was performed in most healthcare settings, this type of education has a short-term impact on patients' attitudes toward self-care activities. a significant gap in primary care about diabetes-related knowledge and practices in caring for patients with diabetes, Previous research has documented a lack of sufficient communication about DSME between patients and physicians.

Diabetes care and education shall be designed with the integration of patient-centered care (PCC), which is a model of clinical practice aimed at shifting patient-provider relationships from authoritarianism to shared decision-making, PCC was described as "providing care that is respectful of and responsive to individual patient preferences, needs, and values and ensuring that patient values guide all clinical decisions".

For enhancing diabetes self-management many educational programs were designed and examined in several studies, the ADA has recommended using the Diabetes self-management education and support (DSMES), which is an education and support model of care designed and provided using a PCC that respects patients' needs and surrounded context with coordination of diabetes nurse and other health care providers efforts, to achieve the seven self-care behaviors of a patient as reliable outcome measures of diabetes self-management " being active, healthy eating, taking medication, monitoring, solving problems, reducing risks and healthy coping" .

Applying the DSMES program produces behavioral changes, empowerment, and cost-effectiveness. In addition, it has a positive impact on health outcomes such as reduces diabetes distress, improves the quality of life, self-efficacy, empowerment, healthy coping, knowledge, and self-care behaviors.

The available evidence suggests that DSME enhance glycemic control but it's not enough alone, many educated patients have well knowledge about diabetes and its management, but they didn't adhere to self-care activities. some literature argues that patients with diabetes need ongoing follow-up and support by diabetes specialists to enhance patients abilities on managing themselves. There have been growing efforts to implement new approaches for self-management interventions that improve diabetes control .

Recently, information technology use has increased dramatically resulting in improved communication. Social Media is defined as the Internet-based tools that permit individuals to communicate, gather and share information, ideas, and images, and to team up with other users in real-time. Social media channels may facilitate digital health interventions, which offer continuous support, efficient communications, and overcome barriers associated with face-to-face modalities. Patients consider social media as a source to get disease-certain information, interact quickly and efficiently with others and share medical information with a community of patients having similar problems.

ELIGIBILITY:
Inclusion Criteria:

1. have a confirmed diagnosis of DM2 in their medical records at last one year.
2. age 18 years old or more
3. able to read and write Arabic
4. agree to participate in the study
5. have uncontrolled blood sugar with HbA1C 8% or more
6. able to use the WhatsApp application
7. Having the ability to autonomous behavior

Exclusion Criteria:

* exclusion criteria:

  1. the presence of mental disorders
  2. complications of acute diabetes or inability to take care of themselves
  3. other serious diseases, such as severe cardiovascular and cerebrovascular diseases, severe kidney disease stage 3, cancer, and visual impairment due to complications of T2DM
  4. gestational diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
glycemic control | baseline and three Monthes post intervention
  This is the primary outcome of the study that will be assessed by the Glycated hemoglobin (A1C)

SECONDARY OUTCOMES:
diabetes self management behaviors | Three moths after the intervention
  will be measured by summary of diabetes self care activities DSCA scale. Is a brief self-report questionnaire and consists of 12 items divided into five self care management activities: diet, practicing exercise, patient self-monitoring of blood glucose, foot care and taking DM medication.This questionnaire is scored by taking the raw score from each set of self care management tasks Then these scores are averaged to form a combined score for each area or subscale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Jordan, Amman, Jordan

REFERENCES:
- [Background] Gabarron E, Arsand E, Wynn R. Social Media Use in Interventions for Diabetes: Rapid Evidence-Based Review. J Med Internet Res. 2018 Aug 10;20(8):e10303. doi: 10.2196/10303. PMID 30097421
- [Background] Zisman-Ilani Y, Obeidat R, Fang L, Hsieh S, Berger Z. Shared Decision Making and Patient-Centered Care in Israel, Jordan, and the United States: Exploratory and Comparative Survey Study of Physician Perceptions. JMIR Form Res. 2020 Aug 3;4(8):e18223. doi: 10.2196/18223. PMID 32744509
- [Result] Ajlouni K, Batieha A, Jaddou H, Khader Y, Abdo N, El-Khateeb M, Hyassat D, Al-Louzi D. Time trends in diabetes mellitus in Jordan between 1994 and 2017. Diabet Med. 2019 Sep;36(9):1176-1182. doi: 10.1111/dme.13894. Epub 2019 Jan 25. PMID 30614070
- [Result] Omar MA, Hasan S, Palaian S, Mahameed S. The impact of a self-management educational program coordinated through WhatsApp on diabetes control. Pharm Pract (Granada). 2020 Apr-Jun;18(2):1841. doi: 10.18549/PharmPract.2020.2.1841. Epub 2020 May 3. PMID 32477434
- [Result] American Association of Diabetes Educators. An Effective Model of Diabetes Care and Education: Revising the AADE7 Self-Care Behaviors(R). Diabetes Educ. 2020 Apr;46(2):139-160. doi: 10.1177/0145721719894903. Epub 2020 Jan 12. PMID 31928334
- [Result] Azami G, Soh KL, Sazlina SG, Salmiah MS, Aazami S, Mozafari M, Taghinejad H. Effect of a Nurse-Led Diabetes Self-Management Education Program on Glycosylated Hemoglobin among Adults with Type 2 Diabetes. J Diabetes Res. 2018 Jul 8;2018:4930157. doi: 10.1155/2018/4930157. eCollection 2018. PMID 30225268
- [Result] Pal K, Dack C, Ross J, Michie S, May C, Stevenson F, Farmer A, Yardley L, Barnard M, Murray E. Digital Health Interventions for Adults With Type 2 Diabetes: Qualitative Study of Patient Perspectives on Diabetes Self-Management Education and Support. J Med Internet Res. 2018 Jan 29;20(2):e40. doi: 10.2196/jmir.8439. PMID 29463488
- [Result] Ventola CL. Social media and health care professionals: benefits, risks, and best practices. P T. 2014 Jul;39(7):491-520. PMID 25083128
- [Derived] Cashmore BA, Cooper TE, Evangelidis NM, Green SC, Lopez-Vargas P, Tunnicliffe DJ. Education programmes for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 Aug 22;8(8):CD007374. doi: 10.1002/14651858.CD007374.pub3. PMID 39171639